CLINICAL TRIAL: NCT00965887
Title: An Open-Label, Randomized, 2-Period Crossover Study to Evaluate the Bioequivalence of a Single Dose of a Tablet Form of MK0974 Ethanolate vs. a Single Dose of a Tablet Form of MK0974 Hydrate in Healthy Subjects
Brief Title: Bioequivalence of Two Tablet Forms of MK0974 (0974-045)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0974-045; MK0974-045; 2009_650
Record Dates: First submitted 2009-08-24; First posted 2009-08-26 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): MK0974 Ethanolate
  Interventions: Drug: MK0974 Ethanolate formulation
- 2 (Active Comparator): MK0974 Hydrate
  Interventions: Drug: Comparator: MK0974 Hydrate formulation

INTERVENTIONS:
Drug: MK0974 Ethanolate formulation — Single dose MK0974 280 mg tablet in one of two treatment periods
  Arms: 1
Drug: Comparator: MK0974 Hydrate formulation — Single dose MK0974 280 mg tablet in one of two treatment periods
  Arms: 2

SUMMARY:
This study will evaluate the bioequivalence of two solid dose formulations of MK0974.

ELIGIBILITY:
Inclusion Criteria:

* Subject is in good health
* Subject is a non-smoker
* Subject is willing to comply with the study restrictions

Exclusion Criteria:

* Subject has a history of stroke, chronic seizures, or major neurological disorder
* Subject has a history of cancer
* Subject is a nursing mother
* Subject has or has a history of any disease or condition that might make participation in the study unsafe or that might confound the results of the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2008-03; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC(0 to infinity) following single dose administration of MK0974 ethanolate or hydrate formulations | Through 48 hours postdose
Peak plasma concentration (Cmax) following single dose administration of MK0974 ethanolate or hydrate formulations | Through 48 Hours Post Dose

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC